CLINICAL TRIAL: NCT00216606
Title: A Randomized Double-Blind Placebo Controlled Trial to Investigate the Efficacy and Tolerability of Topiramate in the Prophylaxis of Chronic Migraine
Brief Title: The Effectiveness and Safety of Topiramate on Prevention of Chronic Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003928
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Migraine
Keywords: Chronic migraine; Migraine; Headache; Migraine headache; Topiramate
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of individualized doses (50 to 200 milligrams) of topiramate tablets compared against placebo for the prevention of chronic migraine headaches over a period of 16 weeks.

DETAILED DESCRIPTION:
Previous studies have shown that topiramate is effective in preventing chronic migraine headaches. This study will start with a 4-week baseline period in which no treatment is given, followed by a 12-week period in which each patient's dose is adjusted and then kept stable for the last 4 weeks of the 16-week double-blind phase. The individualized dose will start at 25 milligrams of topiramate per day and will be increased 25 milligrams per day once weekly and then raised to either the target--100 milligrams per day--or the maximum dose that is well tolerated up to 200 milligrams per day. Patients who are randomized to receive topiramate will remain on the optimized dose. The comparison phase of the study is a 16-week period in which the change in migraine days of patients on topiramate (taking at least 50 milligrams per day) is compared with the change in migraine days for patients on the placebo. Also studied will be the patients' health-related quality of life as assessed by questionnaires filled out at specific visits as well as the patients' views of the safety and tolerability of topiramate. The study hypothesis is that the number of migraine days, periods, and attacks from the baseline period to the last 4 weeks in the double-blind period is reduced more in the topiramate group than the placebo group. During the 16-week comparison period, patients will take by mouth a dose of 50 milligrams to 200 milligrams of topiramate daily.

ELIGIBILITY:
Inclusion Criteria:

* History of migraine for >= 1 year
* Headache type meets HIS (International Headache Society) criteria for migraine
* History reflects "chronic" headache--an average of >= 15 migraine days per month in the 3 months preceding trial entry
* History of chronic migraine for >=1 year>=15 headaches per month with an average duration of 4 hours if not treated
* Patient is otherwise neurologically and physically healthy on a pre-trial exam.

Exclusion Criteria:

* Any other type of chronic headache (besides migraine) from section 2 to 13 of the International Headache Society classification or headache resulting directly resulting some other factor (except for medication overuse)
* Onset of migraine after age 50
* Use of an anticonvulsant drug in the month prior to trial entry
* Use of an antidepressant unless dose has been used at a stable dose for >=3 months
* Use of migraine prevention medicine in the 3 months prior to trial entry unless the drug has been used for at least 3 months and used at a stable dose for at least a month
* Use of a carbonic anhydrase inhibitor such as acetazolamide (used to treat high blood pressure, glaucoma and seizures) or triamterene (a "water pill" for swelling and high blood pressure).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2003-12; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Change in migraine days, migraine periods, and migraine attacks compared between the topiramate group and placebo group at the last month of the baseline phase and the last month of the placebo-controlled phase

SECONDARY OUTCOMES:
Health-related quality of life as recorded in patient questionnaires (MIDAS, HIT-6, MSQ) over 16 double-blind weeks; Patient's satisfaction with the effectiveness and safety of topiramate; Safety

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.